CLINICAL TRIAL: NCT01439464
Title: Clinical Efficacy and Safety of Bioactive Glass-ceramic Intervertebral Spacer (Bonglass-SS) in Posterior Lumbar Interbody Fusion and, Titanium Cage Controlled, 1-year, Single-Blind, Non-Inferiority Trial
Brief Title: Study of Bioactive Glass-ceramic Intervertebral Spacer (Bonglass-SS) in Posterior Lumbar Interbody Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA04-CP01
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Degenerative Disk Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control device (Active Comparator)
  Interventions: Device: 4 CIS one-touch titanium cage
- Investigational device (Experimental)
  Interventions: Device: Bonglass-SS SSLPB

INTERVENTIONS:
Device: 4 CIS one-touch titanium cage — 4 CIS one-touch titanium cage(Solco Biomedical Co. Ltd)
  Arms: Control device
Device: Bonglass-SS SSLPB — Bonglass-SS SSLPB(BioAlpha Inc.)
  Arms: Investigational device

SUMMARY:
The goal of this study is to compare Bonglass-SS with titanum cage.

ELIGIBILITY:
Inclusion Criteria:

* 30~80 aged patients needed single-level posterior Interbody fusion at L1~S1
* A subject who provided written informed consent to participate in this study

Exclusion Criteria:

* Patitents with BMD T-score < -3.0
* Women who are pregnant or plan to be pregnant within 3 years
* Patient with malignant tumor

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessments of fusion and instability at 12 months after surgery | 12 months

SECONDARY OUTCOMES:
CT assessments of fusion at 12 months after surgery | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JaeHyup Lee, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Dongguk University Medical Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Sungnam-Si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Seoul National University Seoul Metropolitan Boramae Medical Center, Seoul